CLINICAL TRIAL: NCT01856725
Title: Evaluation of Programming Strategies for MultiPoint™ Pacing in Cardiac Resynchronization Therapy Patients
Brief Title: MPP Programming Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRD_684
Record Dates: First submitted 2013-05-14; First posted 2013-05-17 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MultiPoint Pacing programming based on hemodynamics (Active Comparator): CRT device implant with MultiPoint Pacing
  Hemodynamic measurements for CRT device programming
  Interventions: Procedure: Hemodynamic measurements for CRT device programming; Device: CRT device implant with MultiPoint Pacing
- MultiPoint Pacing programming without hemodynamics (Experimental): CRT device implant with MultiPoint Pacing
  CRT device programming without hemodynamics
  Interventions: Device: CRT device implant with MultiPoint Pacing

INTERVENTIONS:
Procedure: Hemodynamic measurements for CRT device programming
  Arms: MultiPoint Pacing programming based on hemodynamics
Device: CRT device implant with MultiPoint Pacing

SUMMARY:
The purpose of this study is to compare the efficacy of cardiac resynchronization therapy (CRT) device programming with hemodynamic measurements to device programming without hemodynamic measurements.

ELIGIBILITY:
Inclusion Criteria:

* Be scheduled to undergo implant of a St. Jude Medical (SJM) CRT-D system with approved standard indication by ESC/EHRA Guidelines
* Have the ability to provide informed consent for study participation and be willing and able to comply with the Clinical Investigation Plan (CIP) described evaluations and follow-up schedule

Exclusion Criteria:

* Have high ventricular rate (>90 bpm) during persistent or permanent atrial fibrillation despite available treatment
* Be in NYHA IV functional class
* Have a recent myocardial infarction within 40 days prior to enrollment
* Have undergone cardiac bypass surgery or coronary revascularization procedure within 3 months prior to enrollment or be scheduled for such procedures in the following 7 months
* Have had a recent CVA or TIA within 3 months prior to enrollment
* Have had intravenous inotropic support in the last 30 days
* Be less than 18 years of age
* Be pregnant or planning to become pregnant during the duration of the investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-05; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
end-systolic volume | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Pappone, MD, PhD, Principal Investigator — Maria Cecilia Hospital, GVM Care & Research
Locations (1):
- Maria Cecilia Hospital, GVM Care & Research, Cotignola, RA, Italy